CLINICAL TRIAL: NCT06063941
Title: High-concentration Small-volume Versus Low-concentration Large-volume Iodine Solution for Esophageal Chromoendoscopy: a Multicenter, Randomized Equivalence Trial
Brief Title: High-concentration Small-volume Versus Low-concentration Large-volume Iodine Solution for Esophageal Chromoendoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Collaborators: Ankang Central Hospital (Other); The First Affiliated Hospital of ShiheziI University (Unknown); Xi'an International Medical Center Hospital (Other); Air Force 986 Hospital (Unknown)
Responsible Party: Principal Investigator, Zhiguo Liu, Associate professor, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KY20232274-F-1
Record Dates: First submitted 2023-09-25; First posted 2023-10-03 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Lugol chromoendoscopy; Adverse event
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1% iodine solution arm (Active Comparator): Esophageal chromoendoscopy will be performed with a 15 ml volume of 1% Lugol iodine solution.
  Interventions: Drug: 1% Lugol's iodine solution
- 5% iodine solution arm (Experimental): Esophageal chromoendoscopy will be performed with a 3 ml volume of 5% iodine stock solution.
  Interventions: Drug: 5% Lugol's iodine solution

INTERVENTIONS:
Drug: 1% Lugol's iodine solution — 1% Lugol iodine solution was sprayed from the esophagogastric junction towards a location approximately 20 cm away from the upper incisors in the cervical esophagus.
  Arms: 1% iodine solution arm
Drug: 5% Lugol's iodine solution — Before chromoendoscopy, a 20 ml syringe was employed to draw 3 ml of 5% iodine stock solution and 17 ml air. When staining, the iodine was quickly expelled through the endoscope's working channel at 20 cm of the esophagus from the incisor. An iodine mist was created because of the rapid spurt of the iodine solution and air, which prompts even distribution of the iodine solution on the esophageal wall. The lower segments of the esophageal wall were stained with the remaining iodine solution in the working channel by repeatedly spraying the air/iodine mixture using the syringe, resulting in consistent and uniform staining for the whole esophagus.
  Arms: 5% iodine solution arm

SUMMARY:
This clinical trial aims to test the participants' tolerance for different concentration iodine solutions during esophageal chromoendoscopy. The main question it aims to answer is:

Under the same iodine dosage, do the participants have the same tolerance for 1% and 5% iodine solutions? Participants will be asked to score based on pain and discomfort and describe symptoms and corresponding location at 5 minutes (only for unanesthetized participants) and 30 minutes after chromoendoscopy.

DETAILED DESCRIPTION:
Lugol's iodine chromoendoscopy is the commonly used method for detecting and diagnosing esophageal squamous cell carcinoma. However, iodine can induce mucosal irritation and has been commonly associated with adverse retrosternal symptoms, including retrosternal pain and/or heartburn. The existing research shows that spraying iodine solution neutralizers (Sodium thiosulfate solution, N-acetylcysteine, and vitamin C solution) after esophageal iodine chromoendoscopy can alleviate patient discomfort. However, a recent study has shown that excessive iodine concentration or excessive dosage of iodine can still increase patient discomfort even under spraying an iodine solution neutralizer. It is currently unclear whether the factors affecting patient tolerance are the iodine solution concentration or the total dosage of iodine used. Therefore, the multicenter randomized controlled trial will compare the patient's tolerance for the 1% and 5% iodine solutions under the same iodine dosage conditions. The trial will help determine the specific reasons influencing patient tolerance. Participants will be asked to score based on pain and discomfort and describe symptoms and corresponding location at 5 minutes (only for unanesthetized participants) and 30 minutes after chromoendoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing esophageal Lugol's iodine chromoendoscopy.
* Age ≥ 18

Exclusion Criteria:

* Patients allergic to iodine or with hyperthyroidism;
* Patients with esophageal varices, esophageal ulcer or other conditions inadvisable for Lugol chromoendoscopy;
* Patients with severe gastroesophageal reflux disease or reflux symptoms which may interfered with the outcome measures of current study;
* Patients with postoperative esophageal stenosis affecting endoscopic observation;
* Patients who could not cooperate with the observation and data collection including patients with mental disorders, severe neurosis, dysgnosia or communication disorder;
* Patients with advanced-stage tumors;
* Patients after upper gastrointestinal surgery;
* Patients who do not agree to sign informed consent forms or follow the trial requirement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale scores at 30 minutes after chromoendoscopy | 30 minute after endoscopy
  According to the visual analogue scale, participants will be asked to score based on pain or discomfort 30 minutes after chromoendoscopy.

SECONDARY OUTCOMES:
The color objective evaluation after chromoendoscopy | 2-3 minutes after spraying Lugol's iodine.
  After spraying Lugol's iodine, the esophageal mucosa displaying a homogeneous dark brown staining was classified as normal, while faded or unstained lesions larger than 0.5 cm were deemed potential high-grade intraepithelial neoplasia or mucosal cancer. The Lugol's unstained lesions were further evaluated for the presence of the pink-color sign and photographed 2-3 minutes after Lugol's iodine staining. The images were also taken at 30 cm distal to the incisors at 2-3 minutes after Lugol's iodine staining if no lesion was found. The images were retrospectively analyzed and scored for an objective evaluation based on the L* a* b* (L* = light/dark; a* = red/green; b* = yellow/blue) color values in the CIELAB color space system.
The color subjective evaluation after chromoendoscopy | During endoscopy.
  The endoscopist will be asked to complete a questionnaire survey immediately after chromoendoscopy. The questionnaire asked the endoscopist to rate the staining effect as good (The color concentration is sufficient and the color retention time is adequate) or poor (The color concentration is insufficient and/or the color retention time is inadequate).
Heart rate variability | 5 minute or 30 minute after endoscopy
  The percentage of heart rate change 5 min (only for unanesthetized participants) or 30 min compared to that before endoscopy.
The incidence rate of the need for additional iodine solution spraying | During endoscopy.
  When the endoscopist believes that insufficient esophageal iodine staining affects the detection or diagnosis of lesions, they can spray additional iodine solution. The incidence rate of the need for additional iodine solution spraying of the two groups will be compared.
The dosage of additional iodine spraying | During endoscopy
  When the endoscopist believes that insufficient esophageal iodine staining affects the detection or diagnosis of lesions, they can spray additional iodine solution. The dosage of additional iodine spraying of the two groups will be compared.
Visual analogue scale scores at 5 minutes after chromoendoscopy | 5 minute after endoscopy
  According to the visual analogue scale, participants without sedation or general anesthesia will be asked to score based on pain or discomfort 5 minutes after chromoendoscopy.
The incidence rate of esophageal spasms | During endoscopy
  The incidence rate of esophageal spasms of the two groups will be compared.
The incidence rate of adverse incidents | Up to 48 hours after the endoscopy
  The incidence rate of adverse incidents of the two groups will be compared.
The incidence rate of upper abdominal discomfort or pain. | 5 minute or 30 minute after endoscopy
  Participants will be asked to describe retrosternal discomfort symptoms and corresponding location at 5 minutes (only for unanesthetized participants)) and 30 minutes after chromoendoscopy. The incidence rate of upper abdominal discomfort or pain will be compared between the two groups.
Associated factors for visual analogue scale scores | Up to 48 hours after the endoscopy
  Visual analogue scale scores may be influenced by other factors. Univariable analysis will first be used to identify potential factors that influenced visual analogue scale scores. All possible factors will then be included in multivariable analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiguo Liu, M.D., Principal Investigator — Xijing Hospital of Digestive DIsease
Locations (5):
- China (5):
  - Ankang Central Hospital, Ankang, Shaanxi
  - Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi
  - Air Force 986 Hospital, Xi'an, Shaanxi
  - Xi'an International Medical Center Hospital, Xi'an, Shaanxi
  - The First Affiliated Hospital of Shihezi University, Shihezi, Xinjiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guo Q, Fan X, Zhu S, Zhao X, Fang N, Guo M, Liu Z, Han Y. Comparing N-acetylcysteine with sodium thiosulfate for relieving symptoms caused by Lugol's iodine chromoendoscopy: a randomized, double-blind trial. Gastrointest Endosc. 2022 Feb;95(2):249-257. doi: 10.1016/j.gie.2021.07.025. Epub 2021 Aug 8. PMID 34371004
- [Background] Jin D, Wang J, Zhan Q, Huang K, Wang H, Zhang G, Xu Y, Yao J, Sun R, Huang Q, Ye F, Zhang G. The safety and efficacy of 2% vitamin C solution spray for relief of mucosal irritation caused by Lugol chromoendoscopy: a multicenter, randomized, double-blind, parallel trial. Gastrointest Endosc. 2020 Sep;92(3):554-564. doi: 10.1016/j.gie.2019.11.028. Epub 2019 Nov 26. PMID 31783028
- [Background] Kondo H, Fukuda H, Ono H, Gotoda T, Saito D, Takahiro K, Shirao K, Yamaguchi H, Yoshida S. Sodium thiosulfate solution spray for relief of irritation caused by Lugol's stain in chromoendoscopy. Gastrointest Endosc. 2001 Feb;53(2):199-202. doi: 10.1067/mge.2001.110730. PMID 11174292
- [Background] Liu M, Zhou R, Guo C, Xu R, Liu A, Yang H, Li F, Duan L, Shen L, Wu Q, Liu Z, Liu F, Liu Y, Pan Y, Cai H, Weiss NS, He Z, Ke Y. Size of Lugol-unstained lesions as a predictor for risk of progression in premalignant lesions of the esophagus. Gastrointest Endosc. 2021 May;93(5):1065-1073.e3. doi: 10.1016/j.gie.2020.09.020. Epub 2020 Sep 18. PMID 32950597
- [Background] Park JM, Seok Lee I, Young Kang J, Nyol Paik C, Kyung Cho Y, Woo Kim S, Choi MG, Chung IS. Acute esophageal and gastric injury: complication of Lugol's solution. Scand J Gastroenterol. 2007 Jan;42(1):135-7. doi: 10.1080/00365520600825141. PMID 17190773
- [Background] Tsurumaru D, Utsunomiya T, Matsuura S, Komori M, Kawanami S, Ishibashi T, Honda H. Gastric mucosal changes caused by Lugol's iodine solution spray: endoscopic features of 64 cases on screening esophagogastroduodenoscopy. Gastroenterol Res Pract. 2010;2010:494195. doi: 10.1155/2010/494195. Epub 2010 Apr 12. PMID 20396664
- [Background] Thuler FP, de Paulo GA, Ferrari AP. Chemical esophagitis after chromoendoscopy with Lugol's solution for esophageal cancer: case report. Gastrointest Endosc. 2004 Jun;59(7):925-6. doi: 10.1016/s0016-5107(04)00173-7. No abstract available. PMID 15173818
- [Background] Gotoda T, Kanzaki H, Okamoto Y, Obayashi Y, Baba Y, Hamada K, Sakae H, Abe M, Iwamuro M, Kawano S, Kawahara Y, Okada H. Tolerability and efficacy of the concentration of iodine solution during esophageal chromoendoscopy: a double-blind randomized controlled trial. Gastrointest Endosc. 2020 Apr;91(4):763-770. doi: 10.1016/j.gie.2019.10.022. Epub 2019 Oct 25. PMID 31669091